CLINICAL TRIAL: NCT00272246
Title: Bilateral Internal Pallidum Stimulation in Primary Generalized Dystonia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Princess Beatrix Muscle Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DYSPAS
Record Dates: First submitted 2006-01-04; First posted 2006-01-05 (Estimated); Last update posted 2006-01-05 (Estimated); Status verified 2006-01

CONDITIONS: Dystonia; Primary Generalized Dystonia
Keywords: dystonia
MeSH Terms: conditions — Dystonia

INTERVENTIONS:
Procedure: deep brain stimulation of the internal globus pallidus

SUMMARY:
Primary generalized dystonia, also called idiopathic torsion dystonia or dystonia musculorum deformans is a disabling neurological condition which usually starts in childhood, mostly in a lower limb and spreads to other body parts as the disease progresses. Medical treatment is usually ineffective and most patients become wheelchair bound or even bedridden. Recently several case series and one RCT reported favourable results of bilateral deep brain stimulation (DBS) of the globus pallidus internus (GPi) for primary generalized dystonias. However, the number of patients treated with bilateral GPi stimulation is still limited. Therefore, we propose a RCT to investigate whether bilateral DBS of the GPi is an effective and safe treatment in patients with primary generalized dystonia.

DETAILED DESCRIPTION:
Study design and methods:

This is a randomised, double-blind, placebo-controlled, multicentre study comparing the effect of bilateral DBS of the GPi with placebo in patients with invalidating primary generalized dystonia. After inclusion in the study (see in/exclusioncriteria), a preoperative formal baseline assessment is performed. Within six weeks after the inclusion the patients undergo the stereotactic implantation of the stimulation equipment in the GPi. Immediately after surgery the patients are randomly allocated to direct stimulation (treatment group) or delayed stimulation (control group), in which the stimulator will se switched on 0 Volt before discharge from the hospital by an independent neurologist or neurosurgeon. The patients in both groups are able to control whether the stimulation is active (>0 Volt) or not. In this way the patients and the assessors are blinded. In each centre the postoperative care of the patients will take place according to a stratified stimulation parameter protocol which assures comparable information in both groups. Six months postoperatively, the first formal outcome assessment is performed by the same blinded assessor. After completion of this assessment the stimulators in the control group are activated by an independent neurologist or neurosurgeon. From this moment, all 24 patients have active DBS. However, the patients and blinded assessor remain unaware of the result of the randomisation. All patients are followed for another six months after which the second outcome assessment is made by the same assessor. Four Dutch centres experienced in DBS have agreed to participate in the study. It is estimated that each centre will include at least 4 patients. Because these centra are geographically spread over the country patients can be operated and controlled nearby.

ELIGIBILITY:
Inclusion Criteria:

1. Invalidating primary generalized dystonia (BFMDRS-motor part >= 35)
2. Disease duration >= 5 yrs
3. Age at surgery between 12 and 60
4. Insufficient improvement with pharmacological and physical therapy
5. Signed informed consent, for patients < 19 yrs of age a written consent of the parent(s) or caretaker(s) is needed.

Exclusion Criteria:

1. Mental retardation or dementia (MMSE <24)
2. Depressive state (HADS>21)
3. History of former stereotactic brain surgery
4. Severe brain atrophy
5. General surgical contraindications, such as uncontrolled hypertension or diabetes mellitus, cardiovascular or pulmonary risks, disturbances of bloodclotting.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24
Dates: Start 2005-02; Study Completion 2007-12

PRIMARY OUTCOMES:
change in BFMDRS-motor score from baseline to six months after stimulation equipment implantation

SECONDARY OUTCOMES:
BFMDRS-disability score
MOS-SF-36 (Medical Outcome Scale)
GOS (Global Outcome Scale)
Neuropsychological and neuropsychiatric validated scales
Questionnaire designed for the registration of the number and extent of morbidity due to the surgical
procedure, stimulation equipment and active stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Hans Speelman, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Department of Neurology, Movement Disorders Center, Amsterdam, Netherlands

REFERENCES:
- [Background] Foncke EM, Speelman JD. [Primary generalized dystonia and deep brain stimulation: a randomized, placebo-controlled, double-blind, multicentre study]. Ned Tijdschr Geneeskd. 2005 May 14;149(20):1123-4. Dutch. PMID 15932141